CLINICAL TRIAL: NCT03860194
Title: Effects of Adequate Dietary Protein With Whey Protein, Leucine, and Vitamin D Supplementation on Sarcopenia in Elderly Subjects：An Open-label, Parallel-group Study
Brief Title: Effects of Dietary Supplements on Sarcopenic Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chih-Chien Lin, Attending physician of the Family Medicine Department, Principal Investigator, Far Eastern Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FarEasternMH105096F
Record Dates: First submitted 2019-01-28; First posted 2019-03-01 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supp group (Experimental): Each participant received nutritional counseling and recommended each of them to consume 1.5 g protein/kg body weight (BW)/day. Participants were encouraged to consume a balanced diet with six food groups follow "Daily dietary guideline of 2013 " as recommended by the Ministry of Health and Welfare of Taiwan. However, 1.2 g protein/kg body weight (BW)/day was suggested from this guideline.
  Subjects in the Supp group were provided with Protison with High Protein 51(Original Flavor) containing supplements in addition to their regular daily meals to achieve 1.5 g protein/kg (BW)/day on the basis of this guideline.
  Interventions: Dietary Supplement: Protison with High Protein 51(Original Flavor)
- Diet group (No Intervention): Each participant received nutritional counseling and recommended each of them to consume 1.5 g protein/kg body weight (BW)/day. Participants were encouraged to consume a balanced diet with six food groups follow "Daily dietary guideline of 2013 " as recommended by the Ministry of Health and Welfare of Taiwan. However, 1.2 g protein/kg body weight (BW)/day was suggested from this guideline.
  Subjects in the Diet group were instructed to consume ordinary high protein foods to achieve 1.5 g protein/kg body weight (BW)/day on the basis of this guideline, and suggested to equally distribute their meal time.

INTERVENTIONS:
Dietary Supplement: Protison with High Protein 51(Original Flavor) — Contents of each supplement sachet has a calorie of 88 kcal, 12.8 g protein( including 8.5 g whey protein concentrate), 1.2 g leucine, 7.3 g carbohydrates, 0.8 g fat and 120 IU vitamin D per serving. This supplement was added 200 ml water and stirred well, then drank before meal.
  Arms: Supp group

SUMMARY:
Sarcopenia is defined as a syndrome characterized by decline of skeletal muscle mass and strength or an alteration in physical function. Although some studies showed nutritional supplementation alone might have health benefits for older sarcopenic patients, the results were inconsistent and remain controversial. The objective of this study was to evaluate if a sufficient protein diet including supplements with leucine-enriched whey protein and vitamin D can lead to better improvement than sufficient dietary protein alone in maintaining muscle mass and strength among sarcopenic elders.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (≥ 65 years)
* Subject has lower appendicular muscle mass index (AMMI) (<7 kg/m^2 in men; <5.7 kg/m^2 in women) using Bioelectrical impedance analysis (BIA, TANITA BC-418®, Tokyo, Japan)
* Subject has lower handgrip strength (<26 kg in men; <18 kg in women) using dynamometer (CAMRY®, Zhongshan, Guangdong) or slowly gait speed (<1 m/s)

Exclusion Criteria:

* Subject's life expectancy was shorter than 6 months
* Nursing home resident
* Subject has the history of kidney failure
* Subject has the history of liver failure
* Subject has the history of diabetes mellitus
* Subject has resistance exercise habit.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
AMMI(appendicular muscle mass index) | Change measures (baseline and 4 weeks, baseline and 12 weeks)
  Bioelectrical impedance analysis was used to obtain appendicular muscle mass (AMM) and height. The unit of AMM and height were represented as kilogram and meter respectively. AMMI were calculated as AMM/height^2 (kg/m^2).
Handgrip strength | Change measures (baseline and 4 weeks, baseline and 12 weeks)
  Hand dynamometer was used to measure handgrip strength. Subject was asked to sit in an upright position with the upper arm forming a virtually 90 degree angle with the forearm. Three consecutive measurements of grip strength obtained from both hands were recorded and average of the highest value was calculated as the maximum grip strength. The unit of handgrip strength was represented as kilogram.
Gait speed | Change measures (baseline and 4 weeks, baseline and 12 weeks)
  Asking the subjects to perform a 5-meter walk at their usual pace and measure how much second they could complete this distance, then the unit of gait speed was represented as m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chien Lin, Study Chair — Family Medicine department
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Banciao Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Lin CC, Yeh SL. Reply to the letter to the editor: Effects of adequate dietary protein with whey protein, leucine, and vitamin D supplementation on sarcopenia in older adults: An open-label, parallel-group study. Clin Nutr. 2022 Mar;41(3):792-793. doi: 10.1016/j.clnu.2022.01.030. Epub 2022 Feb 5. PMID 35177293
- [Derived] Lin CC, Shih MH, Chen CD, Yeh SL. Effects of adequate dietary protein with whey protein, leucine, and vitamin D supplementation on sarcopenia in older adults: An open-label, parallel-group study. Clin Nutr. 2021 Mar;40(3):1323-1329. doi: 10.1016/j.clnu.2020.08.017. Epub 2020 Aug 27. PMID 32928579